CLINICAL TRIAL: NCT04764643
Title: The Efficacy of N-acetylcysteine on Alleviating Symptom Caused by Lugol Chromoendoscopy: a Prospective, Non-inferiority, Randomized Controlled Trial
Brief Title: The Efficacy of N-acetylcysteine on Alleviating Symptom Caused by Lugol Chromoendoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KY20202056-F-1
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: lugol chromoendoscopy; adverse event
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium thiosulfate solution arm (Active Comparator): 20ml of 5% sodium thiosulfate solution were prepared with 1g sodium thiosulfate crystal dissolved in normal saline in a 20 ml syringe
  Interventions: Drug: sodium thiosulfate solution
- N-acetylcysteine solution arm (Experimental): 20ml of 3% N-acetylcysteine solution were prepared with one piece of N-acetylcysteine effervescent tablet （ net weight 0.6g ）dissolved in normal saline in a 20 ml syringe
  Interventions: Drug: N-acetylcysteine solution

INTERVENTIONS:
Drug: N-acetylcysteine solution — use N-acetylcysteine solution to alleviate esophageal irritation caused by Lugol's chromoendoscopy
  Arms: N-acetylcysteine solution arm
Drug: sodium thiosulfate solution — use sodium thiosulfate solution to alleviate esophageal irritation caused by Lugol's chromoendoscopy
  Arms: sodium thiosulfate solution arm

SUMMARY:
Lugol chromoendoscopy is essential in detecting and characterizing squamous cell carcinoma of esophagus. Esophageal irritating symptom has been reported as an common adverse event, which could be alleviated by sodium thiosulfate solutions. However, sodium thiosulfate was not widely available. N-acetylcysteine has been previously used as a mucolytic reagent, we propose that it may also be used to alleviate irritating symptoms caused by Lugo's chromoendoscopy. A prospective, non-inferior, randomized double-blind clinical trial was designed to study the efficacy of N-acetylcysteine solutions in relieving esophageal discomfort .

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk of esophageal squamous cell cancer including those over 50 years old, or over 45 years old with family history of esophageal squamous cell cancer;
* Patients with suspected esophageal lesions by screening endoscopy;
* Patients requiring surveillance after endoscopic resection or radiotherapy for esophageal squamous cell cancer one year later。

Exclusion Criteria:

* Patients allergic to iodine or with hyperthyroidism;
* Patients with advanced esophageal cancer, esophageal varices, esophageal ulcer or other conditions inadvisable for Lugol chromoendoscopy;
* Patients with severe gastroesophageal reflux disease or reflux symptoms which may interfered with the outcome measures of current study;
* Patients with postoperative esophageal stenosis affecting endoscopic observation;
* Patients with serious comorbidities that cannot tolerate un-sedated gastroscopy;
* Patients who could not cooperate with the observation including patients with mental disorders, severe neurosis or dysgnosia;
* Patients undergoing sedation or general anesthesia during endoscopy.
* Patients who do not agree to sign informed consent forms or follow the trial requirement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Mean Visual analogue scale change | 30 minute after endoscopy
  Visual analogue scale change for esophageal irritation after Lugol chromoendoscopy

SECONDARY OUTCOMES:
Rate of patients with symptom | 5 minute or 30 minute or 24 hour after endoscopy
  The percentage of patients with symptom after Lugol chromoendoscopy for certain time
Neutralization rate | During endoscopy
  Neutralizing effect for residual iodine in esophagus and stomach
Heart rate variability | 5 minute or 30 minute after endoscopy
  the percentage of heart rate change 5 min or 30 min compared to that Before endoscopy
Severe discomfort rate | 5 minute or 30 minute after endoscopy
  the percentage of patient with Visual analogue scale over 4
exam time | during endoscopy
  the time of endoscopy from the beginning of spraying diluted Lugol's solution to end of endoscopy minus time required for biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Zhu, Principal Investigator — Xijing Hospital of Digestive DIsease
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Kondo H, Fukuda H, Ono H, Gotoda T, Saito D, Takahiro K, Shirao K, Yamaguchi H, Yoshida S. Sodium thiosulfate solution spray for relief of irritation caused by Lugol's stain in chromoendoscopy. Gastrointest Endosc. 2001 Feb;53(2):199-202. doi: 10.1067/mge.2001.110730. PMID 11174292
- [Background] Gotoda T, Kanzaki H, Okamoto Y, Obayashi Y, Baba Y, Hamada K, Sakae H, Abe M, Iwamuro M, Kawano S, Kawahara Y, Okada H. Tolerability and efficacy of the concentration of iodine solution during esophageal chromoendoscopy: a double-blind randomized controlled trial. Gastrointest Endosc. 2020 Apr;91(4):763-770. doi: 10.1016/j.gie.2019.10.022. Epub 2019 Oct 25. PMID 31669091
- [Derived] Guo Q, Fan X, Zhu S, Zhao X, Fang N, Guo M, Liu Z, Han Y. Comparing N-acetylcysteine with sodium thiosulfate for relieving symptoms caused by Lugol's iodine chromoendoscopy: a randomized, double-blind trial. Gastrointest Endosc. 2022 Feb;95(2):249-257. doi: 10.1016/j.gie.2021.07.025. Epub 2021 Aug 8. PMID 34371004